CLINICAL TRIAL: NCT06558123
Title: Comparison of the Effects of Single-Level and Two-Level Deep Parasternal Intercostal Plane (DPIP) Block on Postoperative Sternotomy Pain in Cardiac Surgery
Brief Title: Deep Parasternal Intercostal Plane (DPIP) Block
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: istinye university block
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: single level
  Interventions: Procedure: block
- study: two level
  Interventions: Procedure: block

INTERVENTIONS:
Procedure: block — Single Level and Two Level Deep Parasternal Intercostal Plane (DPIP) Block

SUMMARY:
In this study, we aimed to compare the effects of this block, which is routinely applied in our hospital but has not been studied in our hospital or in the literature before, on the pain in the first 24 hours after the operation, between the single-level and the two-level block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* American Society of Anesthesiologists physical status of II-III
* Undergoing elective coronary artery bypass grafting (CABG), valve repair/replacement, or combined CABG/valve procedure via median sternotomy

Exclusion Criteria:

* Patients who are unable to communicate
* Patients who have had emergency surgery, reoperation, thoracotomy or mastectomy
* Patients with a history of chronic pain
* Patients who are using chronic opioids or sedatives
* Patients who have had a re-sternotomy within 24 hours of surgery
* Patients with liver or kidney failure
* Patients who are using narcotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who will undergo sternotomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
numeric rating scale | 4 month
  24 hours pain

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Min J, Chen S. Sensory Assessment and Block Duration of Deep Parasternal Intercostal Plane Block in Patients Undergoing Cardiac Surgery: A Prospective Observational Study. Pain Ther. 2022 Sep;11(3):951-958. doi: 10.1007/s40122-022-00403-y. Epub 2022 Jun 25. PMID 35751781
- [Result] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Result] Gelinas C. Management of pain in cardiac surgery ICU patients: have we improved over time? Intensive Crit Care Nurs. 2007 Oct;23(5):298-303. doi: 10.1016/j.iccn.2007.03.002. Epub 2007 Apr 19. PMID 17448662